CLINICAL TRIAL: NCT06636071
Title: An Open-label Phase 3 Study of Setrusumab in Pediatric Japanese Subjects With Osteogenesis Imperfecta Type I, III, or IV
Brief Title: Setrusumab in Pediatric Japanese Subjects With Osteogenesis Imperfecta
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX143-CL307
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — setrusumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setrusumab (Experimental)
  Interventions: Biological: setrusumab

INTERVENTIONS:
Biological: setrusumab — A fully human sclerostin neutralizing monoclonal antibody (mAb) administered once a month (QM) via intravenous (IV) infusion
  Other Names: BPS804; UX143

SUMMARY:
The primary objective of the study is to evaluate the effect of setrusumab on reduction in fracture rate, including morphometric vertebral fractures.

DETAILED DESCRIPTION:
This study will be conducted in Japan only and consists of a screening period, an open-label treatment period, and an open-label extension period. Participants will receive setrusumab for up to 24 months during the open-label Treatment Period followed by continued setrusumab treatment during the open-label Extension Period. All participants will receive setrusumab until it becomes commercially available in Japan, consent is withdrawn, or the study is otherwise discontinued.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of OI Type I, III, or IV confirmed by identification of genetic mutation in COL1A1 or COL1A2
* History of ≥ 1 fracture in the past 12 months, ≥ 2 fractures in the past 24 months, or ≥ 1 femur, tibia, or humerus fracture in the past 24 months
* Any prior exposure to, or currently receiving, IV-bisphosphonate therapy for treatment of OI
* Serum 25-hydroxyvitamin D level ≥ 20 ng/mL at the Screening visit. If 25- hydroxyvitamin D levels are below 20 ng/mL, the subject may be rescreened after a minimum of 14 days of vitamin D supplementation as directed by the Investigator

Exclusion Criteria:

* History of skeletal malignancies or bone metastases at any time
* History of neural foraminal stenosis (except if due to scoliosis)
* Clinical manifestations of Chiari malformation or basilar invagination. Presence of any other neurologic disease that has been clinically unstable within past 2 years requires review by the Medical Monitor.
* History of or current uncontrolled concomitant diseases that may impact bone metabolism, such as hypo/hyperparathyroidism, abnormal thyroid function, nephrotic syndrome, or Stage IV/V renal disease
* Any skeletal condition (other than OI) leading to bone deformity and/or increased risk of fractures, such as rickets, osteopetrosis, idiopathic juvenile osteoporosis, or skeletal dysplasia
* History of known cardiovascular disease such as coronary artery anomaly, Kawasaki disease, myocarditis, cardiomyopathy, myocardial infarction, stroke, or thromboembolic disease. Individuals with other congenital or acquired cardiovascular disease necessitating an echocardiogram require Medical Monitor review. Investigators should consider whether the potential benefits of treatment outweigh the potential risks in patients with cardiovascular risk factors such as confirmed arterial hypertension.
* Hypocalcemia, defined as serum calcium levels below the age-adjusted normal limit reference ranges after a recommended ≥ 4 hour fast, at Screening
* Estimated glomerular filtration rate ≤ 35 mL/min/1.73 m2 at Screening
* Prior treatment with growth hormone, denosumab, anti-sclerostin antibody, or other anabolic or anti-resorptive medications impacting the bone (other than bisphosphonates) at any time
* History of external radiation therapy
* Known hypersensitivity to setrusumab or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation, pose undue risk, or would confound interpretation of results
* Use of any investigational product or investigational medical device within 4 weeks or 5 half-lives (whichever is longer) of investigational drug prior to Screening, or during the study (per discretion of the Investigator in consultation with the Medical Monitor)
* Concurrent participation in another clinical study without prior approval from the study Medical Monitor
* Pregnant or nursing

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Rate of All Radiographically-Confirmed Fractures, Including Morphometric Vertebral Fractures During the Treatment Period | Up to Month 24

SECONDARY OUTCOMES:
Annualized Rate of Radiographically-Confirmed Fractures, Excluding Morphometric Vertebral Fractures, but Including Fractures of the Fingers, Toes, Face, and Skull During the Treatment Period | Up to Month 24
Annualized Rate of All Radiographically-Confirmed Fractures, Excluding Morphometric Vertebral Fractures and Fractures of the Fingers, Toes, Face, and Skull During the Treatment Period | Up to Month 24
Change from Baseline in Dual-Energy X-Ray Absorptiometry (DXA) Bone Mineral Density (BMD) Z-Score at the Lumbar Spine During the Treatment Period | Baseline, Up to Month 24
Percent Change from Baseline in DXA BMD at the Lumbar Spine During the Treatment Period | Baseline, Up to Month 24
Proportion of Participants Experiencing New Radiographically-Confirmed Fractures, Including Morphometric Vertebral Fractures, at the Primary Analysis | Up to Month 24
Serum Setrusumab Concentration Over Time | Up to Month 24
Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs), Frequency, Severity and Relationship to Treatment | Up to Month 24
Incidence of Binding and Neutralizing Anti-Setrusumab Antibodies Over Time | Baseline, Up to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Ultragenyx Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (3):
- Japan (3):
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Keio University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Osteogenesis Imperfecta (OI) Research Study Opportunity — https://www.ultraclinicaltrials.com/OI
- See also: Our Clinical Trial Transparency Commitment-Ultragenyx — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/